CLINICAL TRIAL: NCT05913817
Title: The Evaluation of Injection Site Pain and Adherence in Patients Switching from a Low to High Concentration Adalimumab (AVT-02) Across Multiple Indications.
Acronym: EASE PAIN
Status: Active, not recruiting | Type: Observational
Sponsor: Jamp Pharma Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: JAMP-AVT02-001
Record Dates: First submitted 2023-06-02; First posted 2023-06-22 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-09

CONDITIONS: Crohn Disease; Ulcerative Colitis; Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis; Plaque Psoriasis; Hidradenitis Suppurativa
Keywords: Injection Site Pain
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Hidradenitis Suppurativa | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adalimumab Reference Product to AVT-02: Patients switching from the high-volume, low concentration, citrate containing Adalimumab reference product to the low-volume, high-concentration, citrate-free AVT-02 Adalimumab Biosimilar.
  Interventions: Biological: AVT02 (Alvotech Biosimilar to Adalimumab)
- Other Adalimumab Biosimilar to AVT-02: Patients switching from another high-volume, low concentration, citrate-containing or citrate-free Adalimumab biosimilar product to the low-volume, high-concentration, citrate-free AVT-02 Adalimumab Biosimilar.
  Interventions: Biological: AVT02 (Alvotech Biosimilar to Adalimumab)

INTERVENTIONS:
Biological: AVT02 (Alvotech Biosimilar to Adalimumab) — Phase IV Study
  Other Names: Humira

SUMMARY:
The purpose of the Phase IV study is to investigate the effects of both Volume and Citrate on Injection Site Pain (ISP), adherence, patient satisfaction, Quality of Life, and Disease Assessment in the Canadian Adalimumab Market.

The phase IV study is an observational, pan-Canadian, multidisciplinary study aiming to enroll 600 patients across 50-70 sites across 3 different Therapeutic Areas (GI, Rheum, Derm).

DETAILED DESCRIPTION:
The current phase 4 study seeks to assess the real-world injection experience, utilization, satisfaction, effectiveness, safety, and tolerability of treatment with AVT-02 (SIMLANDI™) in patients when switching from low-concentration adalimumab Humira® or another adalimumab biosimilar to high-concentration adalimumab SIMLANDI™ for the management of certain gastroenterological (IBD, including CD or UC); rheumatological (including RA, AS, or PsA); or dermatological conditions (including HS or PsO).

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years or older at the time of consent.
2. Patient has been diagnosed with CD, UC, RA, AS, PsA, HS, or PsO for at least 6 months.
3. Patient must be a current user of Humira® or another low-concentration adalimumab biosimilar, with treatment initiated at least 6 months prior to screening.
4. One of the following:

   1. Treating physician is considering switching from Humira® to SIMLANDI™,
   2. Treating physician is considering switching from an adalimumab biosimilar (not Humira®) to SIMLANDI™.
   3. Treating physician has switched from Humira® or Humira® biosimilar to SIMLANDI™ within the past 3 months.
5. Patient must be willing to keep using the same type of injector when switching from their previous adalimumab treatment to SIMLANDI™:

   1. Pre-filled to pre-filled switch,
   2. Autoinjector to autoinjector switch.
6. Access to commercial SIMLANDI™.
7. Patient or patient's legal/authorized representative agrees to sign informed consent and participate in the study.

Exclusion Criteria:

1. Patients previously treated with SIMLANDI™ or another high-concentration adalimumab biosimilar.
2. Patients that, in the opinion of the investigator, have any condition that may impair their ability to participate in the study.
3. Any current or history of any condition that, in the opinion of the investigator, participation in the study may increase the risk to the patient.
4. Patients for whom treatment with adalimumab may be contraindicated (e.g., patients with demyelinating disorders).
5. Patients with moderate to severe heart failure, as indicated by New York Heart Association (NYHA) class >= 3.
6. Patients with severe infections such as sepsis, tuberculosis, or opportunistic infections.
7. Patients with history of recurrent infection or with underlying conditions which may predispose them to infections.
8. Patients with known hypersensitivity to SIMLANDI™ or its excipients.
9. Patients who are unable to secure reimbursement for SIMLANDI™.
10. Patient anticipates not being available for follow-up assessments as required for adequate management.
11. Active participation in or enrollment in an interventional trial.
12. Patient or patient's legal/authorized representative cannot or will not sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To ensure a representative study population, any eligible patient that meets the inclusion/exclusion criteria should be invited to participate in this non-interventional study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-05-13 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in injection site pain after the first dose of high-concentration adalimumab (AVT-02) as measured by the Visual Analog Scale (VAS); 2 weeks after Humira Injection (can be 1 week for certain indications such as HS). | At 2 Weeks
  Baseline injection site pain will be defined as the VAS score recorded during the last dose of the low-concentration adalimumab prior to switching to AVT-02.

SECONDARY OUTCOMES:
Change from baseline in injection site pain after every injection of the high-concentration adalimumab (AVT-02) as measured by VAS during the 180 days of the study. | At Every AVT-02 Injection up to 180 Days.
  Baseline injection site pain will be defined as the VAS score recorded during the last dose of the low-concentration adalimumab prior to switching to AVT-02.
Patient perception of change in injection site pain (5-point Likert) after the first dose of high-concentration adalimumab (AVT-02) compared to Humira® or another low-concentration adalimumab biosimilar. | Once a month up to 180 Days.
  A five-point Likert scale of patient perception of change in injection site pain after the first dose of high-concentration adalimumab (AVT-02).
Distribution of missed doses of AVT-02. | At Every AVT-02 Injection up to 180 Days.
  Adherence to treatment when switching from Humira® or another adalimumab biosimilar to AVT-02.
Change from baseline in overall satisfaction with the injection (7-point Likert) during the 180 days of the study after switching from Humira or another low-concentration adalimumab to AVT-02. | At Every AVT-02 Injection up to 180 Days.
  A seven-point Likert scale of patient satisfaction.
Change from baseline in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Index Score during the 180 days of the study after switching from Humira or another low-concentration adalimumab to AVT-02. | At days 30, 60, 90, 120, 150, and 180.
  A questionnaire assessing health-related quality of life covering five dimensions (mobility, ability to self-care, ability to undertake usual activities, pain/discomfort, and anxiety/depression) with five levels of severity for each dimension (no problems, slight problems, moderate problems, severe problems, and extreme problems).
Change from baseline in physician disease assessment during the 180 days of the study after switching from Humira or another low-concentration adalimumab to AVT-02 | At Baseline and at Day 180.
  Asses the Physician Global Assessment (PGA) at baseline and at Day 180.
Change from baseline in patient-reported disease assessment during the 180 days of the study after switching from Humira or another low-concentration adalimumab to AVT-02 | At Baseline and at Day 180.
  Asses the Patient Global Assessment of Disease Activity (PtGA) at baseline and at Day 180.
Change from baseline in health care utilization during the 180 days of the study. | At days 30, 60, 90, 120, 150, and 180.
  A questionnaire assessing healthcare resource utilization related to the patient indication, including medical events and treatments experienced by the patient in the last month.

CONTACTS AND LOCATIONS:
Locations (1):
- JAMP Pharma Corporation, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No